CLINICAL TRIAL: NCT00484614
Title: Prospective Multicenter Study of the Role of Positron Emission Mammography (PEM) in Pre-Surgical Planning for Breast Cancer
Brief Title: Study the Role of Positron Emission Mammography in Pre-surgical Planning for Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Naviscan PET Systems (Industry)
Collaborators: Certus International, Inc. (Other)
Responsible Party: Judith E Kalinyak, Medical Director, Naviscan PET Systems, Inc
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: PEM-06-01; NIH Grant: 5 R44 CA103102-05
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2008-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer, breast conserving surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 PEM (Active Comparator)
  Interventions: Procedure: Positron Emission Mammography
- 2 MRI (Active Comparator)
  Interventions: Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Positron Emission Mammography — Molecular Imaging Device
  Other Names: Naviscan PET Systems, PEM Flex Solo
  Arms: 1 PEM
Procedure: Magnetic Resonance Imaging — Imaging Device
  Arms: 2 MRI

SUMMARY:
Women with newly diagnosed breast cancer anticipating breast-conserving surgery are enrolled into the study and will undergo both high-resolution positron emission mammographic (PEM) imaging and contrast-enhanced magnetic resonance imaging (MRI) of the breast(s). The purpose of this study is to determine changes in surgical management resulting from PEM or MRI imaging as compared to conventional imaging and to determine if the changes were appropriate with histopathology as gold standard.

DETAILED DESCRIPTION:
Breast compression and/or immobilization during positron emission tomographic (PET) imaging has been called positron emission mammography, or "PEM," and the device used to perform the scan has been called a PEM Scanner. This protocol is designed as a prospective multi-center clinical trial to evaluate the role of high resolution PEM, used in combination with the radiotracer 2-[F-18]- fluorodeoxyglucose (FDG), in pre-surgical planning in women with newly diagnosed breast cancer who are considered candidates for breast conserving surgery (i.e. lumpectomy) after full workup with mammography, clinical breast exam, and additional US as would normally be performed. Participants will undergo both contrast enhanced MRI and PEM imaging. In order to control for potential bias in interpretation of the second examination (i.e. PEM or MRI), the order of interpretation of these examinations will be randomly assigned at study entry.The primary objective of the study is to determine changes in surgical management resulting from PEM or MRI or both, separately and in conjunction with conventional imaging and to determine whether these changes were appropriate (i.e. to excise malignancy) or inappropriate (e.g. wider excision or mastectomy for what proved to be benign disease).

ELIGIBILITY:
Inclusion Criteria:

1. Women who are 25 years of age or older
2. Newly diagnosed core-biopsy proven breast cancer
3. Has current mammography of all study breasts (within prior 3 months), including magnification views of suspicious calcifications (if any)
4. Recent clinical breast examination (within prior 3 months)
5. Has had full diagnostic workup with breast ultrasound (within prior 3 months) as indicated by mammographic and/or clinical findings
6. Has had percutaneous biopsy of all relevant suspicious findings on mammography, clinical examination, and ultrasound
7. After full diagnostic workup, participant is likely to be a candidate for breast conserving surgery.
8. No contraindications to breast MRI:

   * No pacemaker, aneurysm clip, or other implanted magnetic or ferromagnetic device;
   * No claustrophobia that cannot be controlled by medication with valium, ativan, or other sedative under her physician's orders;
   * Has intravenous access;
   * Weight < 300 lbs;
   * Physically able to tolerate positioning in the MRI scanner.
9. Agrees to undergo follow-up MRI or PEM at 6 months and/or MRI-guided vacuum-assisted biopsy, US-guided core biopsy, or PEM-guided biopsy if needed based on results of the MRI or PEM examination
10. Has signed study-specific consent form
11. Subject agrees to undergo a contrast-enhanced MRI and PEM scan within five business days of each other, prior to surgery.

Exclusion Criteria:

1. Male
2. Pregnancy
3. Active lactation or discontinued breastfeeding < 2 months prior
4. Age less than 25 years
5. Inability to provide informed consent
6. Prior radiation treatment to the affected breast(s)
7. Participant is scheduled for sentinel node procedure using radioactive Tc-99m within 24 hours after the scheduled PEM Flex study
8. Women planning prophylactic mastectomy without histologic confirmation
9. Individuals who are electing to undergo neoadjuvant chemotherapy prior to surgery (Note: Patients with prior contralateral breast cancer receiving chemoprevention with Tamoxifen, Arimidex, or other aromatase inhibitor are eligible)
10. Individuals who have had surgery on the study breast(s) within the past 12 months
11. Breast implant(s) in any study breast(s)
12. Women who have had distant metastatic disease either currently or in the past
13. Individuals with Type I or poorly controlled Type II diabetes mellitus
14. Individuals with a blood glucose level that is above 140 mg/dl at the time of PEM imaging
15. Has not had contrast-enhanced breast MRI or PEM within the past 12 months prior to study enrollment
16. Subject is currently enrolled in another breast imaging research study

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2006-09; Primary Completion 2008-11 (Actual); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
The primary outcome for this study will be measured by evidence of malignancy on PEM and/or MRI, confirmed by core biopsy or surgery. | Within 30 days (plus or minus a week) after core biopsy/surgery

SECONDARY OUTCOMES:
Risk of false positive examinations with either PEM or MRI imaging with surgery as gold standard | Within the first 30 days (plus or minus 7 days) after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wendie A Berg, MD, Ph.D, Study Director — American Radiology Services, Johns Hopkins Greenspring, Lutherville, MD; Etta Pisano, MD, FACR, Principal Investigator — University of North Carolina School of Medicine, Chapel Hill, NC; Kathy Schilling, MD, Principal Investigator — Boca Raton Community Hospital, Boca Raton, FL; Marie Tartar, MD, Principal Investigator — Scripps Cancer Center, San Diego, CA; Linda Hovanessian Larsen, MD, Principal Investigator — USC Norris Cancer Center; Lorraine Tafra, MD, Principal Investigator — Anne Arundel Medical Center, MD
Locations (6):
- United States (6):
  - University of Southern California, Los Angeles, California
  - Scripps Cancer Center, San Diego, California
  - Boca Raton Community Hospital, Boca Raton, Florida
  - Anne Arundel Medical Center, Annapolis, Maryland
  - American Radiology Services, Inc., Johns Hopkins Green Spring, Lutherville, Maryland
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina

REFERENCES:
- [Background] Berg WA, Weinberg IN, Narayanan D, Lobrano ME, Ross E, Amodei L, Tafra L, Adler LP, Uddo J, Stein W 3rd, Levine EA; Positron Emission Mammography Working Group. High-resolution fluorodeoxyglucose positron emission tomography with compression ("positron emission mammography") is highly accurate in depicting primary breast cancer. Breast J. 2006 Jul-Aug;12(4):309-23. doi: 10.1111/j.1075-122X.2006.00269.x. PMID 16848840
- [Background] Tafra L, Cheng Z, Uddo J, Lobrano MB, Stein W, Berg WA, Levine E, Weinberg IN, Narayanan D, Ross E, Beylin D, Yarnall S, Keen R, Sawyer K, Van Geffen J, Freimanis RL, Staab E, Adler LP, Lovelace J, Shen P, Stewart J, Dolinsky S. Pilot clinical trial of 18F-fluorodeoxyglucose positron-emission mammography in the surgical management of breast cancer. Am J Surg. 2005 Oct;190(4):628-32. doi: 10.1016/j.amjsurg.2005.06.029. PMID 16164937
- See also: Sponsor's website — http://www.naviscanpet.com